CLINICAL TRIAL: NCT05388201
Title: Variation In Facial Morphology As A Determinant Of Face Covering Performance: FACEFIT
Acronym: FACEFIT
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 20-2612
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: Healthy Subjects; Mask; Mask Fit; Fitted Filtration Efficiency; Facial Features; Craniofacial Morphology; 3D Facial Imaging; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — N95 Respirators; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FACEFIT: Participants will enter a chamber where they will undergo 3D facial scanning using a dedicated camera system and be trained to don a N95 respirator properly. The fitted filtering efficiency (FFE) of 4 types of face coverings: a N95 respirator, a KN95 respirator (with and without a clip), a surgical mask (with and without a clip), and a KF94 respirator (with and without a clip) will be tested using the OSHA quantitative fit testing protocol for filtering face pieces. Participants will measure their peak expiratory flow pre and post mask fit testing using a disposable peak flow meter.
  Interventions: Other: N95; Other: KN95; Other: KF94; Other: Surgical

INTERVENTIONS:
Other: N95 — 3M N95 Respirator
Other: KN95 — KN95 Mask (with and without clip)
Other: KF94 — KF94 Mask (with and without clip)
Other: Surgical — Surgical Mask (with and without clip)

SUMMARY:
This study examines the role of variations in the dimensions of facial features on the fitted filtering efficiency of face coverings available to the public during the COVID-19 pandemic. Approximately 100 young (18-55 years old) healthy participants will be recruited. Exclusionary criteria include pregnancy and breastfeeding. After informed consent, participants will enter a chamber where they will undergo 3D facial scanning using a dedicated camera system and be trained to don an N95 respirator properly. The fitted filtering efficiency (FFE) of 4 types of face coverings: a N95 respirator, a KN95 respirator (with and without a clip), a surgical mask (with and without a clip), and a KF94 respirator (with and without a clip) will be tested on each participant using the OSHA quantitative fit testing protocol for filtering face pieces.

DETAILED DESCRIPTION:
Consenting: The investigators will review the inclusion and exclusion criteria and any medical conditions that the participant may have or medications that they are currently taking. The investigators will go over the study protocol in detail so that the participant will know what to expect during the study procedure.

Lung Function Test: The participant will perform a breathing test (peak flow meter) before and after the facemask testing. This test measures the volume of air that the participant can blow out (exhale) quickly after taking a very deep breath. This is a method for measuring lung function and it must meet certain criteria prior to testing.

3D Facial Measurement and Imaging: The participants 3D facial features will be measured by facial calipers. Trained personnel (wearing gloves) will need to touch areas of the participants face and scalp to ensure proper caliper measurements are collected. A 3D picture of the participants face will be taken using a special 3D camera.

Video Instruction on Wearing an N-95 Respirator: The participant will watch a short video showing proper ways to wear an N-95 respirator.

Assessment of the Performance of Face Coverings: The participant will enter a study chamber where tiny sodium chloride (table salt) particles are emitted by a particle generator. The participant will be fit tested wearing different types of face coverings that include an N95-rated respirator, a KN95 mask (with and without clip), a surgical mask (with and without clip), and a KF94 respirator (with and without clip). During the test, the participant will be asked to perform a few tasks such as bending over, talking, etc. 3D images of the participants head, while wearing the masks, will be taken following each test.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years old healthy male and female (BMI values between 19 and 33, inclusive).
* Participants must be ambulatory and tolerate enclosed spaces.
* Participants must be up to date with their COVID-19 vaccination status based on the current recommendations established by the CDC.

Exclusion Criteria:

* Individuals with following conditions:

  * A history of acute or chronic cardiovascular disease, chronic respiratory disease, cancer, rheumatologic disease, neuromuscular disease, or immunodeficiency state.
  * Blood pressure readings equal to and greater than 140 systolic and equal to and greater than 90 diastolic.
  * Diabetes.
  * Asthma or a history of asthma.
* Individuals who have unspecified illnesses, which in the judgment of the medical staff might increase the risk associated with saline aerosol inhalation will be a basis for exclusion.
* Medications not specifically mentioned here may be reviewed by the medical staff prior to an individual's inclusion in the study. Use of other medications will be evaluated on a case-by-case basis. There is the potential that an individual's current medication use will preclude them from participating in the study at the current time, but they may be reassessed and potentially rescheduled for participation later based on the judgement of the medical staff.
* Individuals who are pregnant, attempting to become pregnant or breastfeeding.
* Individuals who are currently smoking (including vaping, hookah and e-cigarette) or have smoking history within 1 year of study or have a greater than/equal to a 5-pack year smoking history.
* Individuals living with a smoker who smokes inside the house.
* Individuals who are regularly exposed to high levels of vapors, dust, gases, or fumes.
* Individuals who do not read, speak, or understand English well enough to give informed consent.
* Individuals who are unwilling to shave facial hair.
* Individuals who have orthopedic or balance issues that prevent them from performing the steps in the mask fit testing protocol, such as bending over, turning head left and right or up and down.
* Individuals who recently had abdominal and/or eye surgery, or with any types of hernia, as well as any other contraindications for raised intra-abdominal pressure in the last 6 months.

Temporary exclusion criteria:

* Individuals who have experienced any symptoms associated with acute respiratory illness within 4 weeks of enrollment.
* Individuals who have active allergies.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male and female subjects
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Fitted Filtration Efficiency (FFE) | Approximately 5 minutes after each mask condition
  A mask fit procedure will be performed based on a NIOSH (National Institute of Occupational Safety and Health) - approved protocol during the baseline visit. The efficiency of masks will be determined by a percentage of particle number measured behind the facemask over the particle number in the ambient air. Mask fit efficiency values from different levels of mask fit instructions will be compared.
Craniofacial Morphology | Approximately 5 minutes before mask donning
  Calipers will be used to measure 3D facial features of each subject. Trained personnel (wearing gloves) will need to touch areas of the subject's face and scalp to ensure proper caliper measurements are collected.

SECONDARY OUTCOMES:
3D Facial Imaging | Approximately 5 minutes before mask donning and during mask donning
  Subjects will self-administer a 3D scan of their face by aligning their head inside of an oval shown on the camera screen, triggering the camera shutter. The image takes about 3 seconds to generate and subjects will be asked to remain still during this time. The acquired facial images will be analyzed using digital image analysis software.

CONTACTS AND LOCATIONS:
Overall Officials: James Samet, PhD, Principal Investigator — Environmental Protection Agency (EPA)
Locations (1):
- U.S. Environmental Protection Agency Human Studies Facility, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data will be shared through the U.S. EPA's ScienceHub database. ScienceHub is used to upload and store datasets associated with journal articles. Non-sensitive datasets are then made publicly accessible via the Environmental Dataset Gateway in fulfillment of the EPA's requirement to adhere to the Office of Management and Budget's Open Data Policy.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available to the public after the conclusion of the study and the publication of the manuscripts.
Access Criteria: Data will be available at the U.S. EPA Science Hub.
URL: https://catalog.data.gov/dataset/epa-sciencehub

REFERENCES:
- [Derived] Griffin JS, McInroe EM, Pennington ER, Steinhardt W, Chen H, Prince SE, Samet JM. Craniometric determinants of the fitted filtration efficiency of disposable masks. Front Public Health. 2024 Aug 20;12:1444411. doi: 10.3389/fpubh.2024.1444411. eCollection 2024. PMID 39228845